CLINICAL TRIAL: NCT06997653
Title: Open-Label, Phase 2b Clinical Trial to Determine Efficacy, Safety, and Immunogenicity of Inactivated COVID-19 Vaccine (TURKOVAC) Against SARS-CoV-2 in Healthy Pregnant Women
Brief Title: Efficacy, Immunogenicity, and Safety of the Inactivated COVID-19 Vaccine (TURKOVAC) in Healthy Pregnant Women
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the clinical trial did not initiated
Sponsor: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TBS-VAC-COV-TUR-GF2B.08
Record Dates: First submitted 2022-03-09; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: COVID-19; SARS CoV 2 Infection
Keywords: COVID-19; SARS-CoV-2 Vaccine; Pregnant Women; Efficacy; Immunogenicity; Safety
MeSH Terms: conditions — COVID-19 | interventions — TURKOVAC

STUDY DESIGN:
Masking Description: Open-Label, National, Phase IIB Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TURKOVAC (Experimental): TURKOVAC-Dollvet vaccines produced by Dollvet Veterinary Vaccine Pharmaceutical Biological Substance Production Industry Co., Ltd.
  Interventions: Biological: TURKOVAC

INTERVENTIONS:
Biological: TURKOVAC — Inactive COVID-19 Vaccine - TURKOVAC

SUMMARY:
This study is an open-label and Phase 2b clinical trial of the COVID-19 inactivated TURKOVAC vaccine against SARS-CoV-2 in healthy pregnant women.

DETAILED DESCRIPTION:
The main purpose of this study is pregnant women who are at least in the second (13th to 27th weeks) and third (28th to 40th weeks) trimesters, to evaluate of the safety of two doses of TURKOVAC vaccine in who are naive (never vaccinated) and previously vaccinated with two doses of inactivated COVID-19 vaccine.

It is planned to include 30 healthy pregnant subjects between the ages of 18-45 (including both age groups) in the study. After the safety and immunogenicity data obtained from the interim analysis of 30 pregnant female subjects, it will be planned to increase the number of subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Subjects willing and able to give signed informed consent to participate in study,
2. Healthy pregnant female subjects aged 18 - 45 years (including both groups),
3. Females in the second trimester of pregnancy (weeks 13 to 27) and in the third trimester (from week 28 to week 40),
4. Females who were previously vaccinated with two doses of inactivated vaccine also 3 months after their last menstrual period and more than 3 months have passed since they have vaccinated for their last dose,
5. Females without a current positive (real time-polymerase chain reaction (RT-PCR) - based viral RNA (Ribonucleic Acid) detection) or past (serological test or real time-polymerase chain reaction (RT-PCR -based viral RNA (Ribonucleic Acid) detection) positive diagnostic test result for SARS-CoV-2 infection,
6. In the opinion of the investigator, subjects capable and willing to comply with all study requirements,
7. Subjects who agree to comply with all study visits and procedures (who consent to blood and nasopharyngeal swab collection and who can answer automated phone calls from the study center).

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Subjects with fever (above 37,8°C) at the time of vaccination and/or up to 72 hours before (subjects may be screened again after acute condition has resolved),
2. Possible history of allergic disease or reaction (e.g. to the active substance) by any component of the study vaccines,
3. Any history of anaphylaxis,
4. Subjects with a medical or obstetric history that puts them at higher risk for maternal or fetal complications (e.g. chronic pregnancy-related disorders, birth defects, or genetic conditions during a previous pregnancy),
5. Subjects with an abnormal uterine cavity shown on hysterosalpingography or hysteroscopy,
6. Subjects with an abnormal pregnancy screening test (e.g. ultrasound fetal abnormalities, maternal blood screening),
7. Subjects with a history of malignancy within 2 years prior to screening (exceptions are squamous, basal cell carcinomas of the skin, carcinomas in situ of the cervix, or malignancy considered treated with minimal risk of recurrence),
8. Females with the presence of hydrosalpinx or endometrial polyp that are not treated surgically,
9. Females with the poor ovarian response (less than 3 mature follicles),
10. Females currently participating in a similar study of another inactive investigational product and currently using this investigational product or who have taken an inactive investigational product in the 28 days before their last menstruation period,
11. In case of clinical necessity, subjects with positive COVID-19 real time-polymerase chain reaction (RT-PCR) test results to be requested from the subjects,
12. Insufficient level of Turkish to perform the informed consent, except where briefing by an independent witness can be provided and is available,
13. Any other significant disease, disorder or finding that could significantly increase the subject's risk for participation in the study, affect the subject's ability to participate in the study, or impair the interpretation of study data; severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, kidney disease, endocrine disorder, and neurological disease (mild/moderate well-controlled comorbidities are permitted),
14. Any confirmed or suspected immunosuppressive or immunodeficiency state; asplenia; recurrent severe infections and use of immunosuppressants (less than ≤14 days) in the last 6 months, excluding topical steroids or short-term oral steroids,
15. History of bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venipuncture,
16. Continued use of anticoagulants such as coumarins and related anticoagulants (e.g. warfarin) or new oral anticoagulants (e.g. apixaban, rivaroxaban, dabigatran and edoxaban),
17. Subjects with cerebral venous sinus thrombosis, antiphospholipid syndrome, or a history of heparin-induced thrombocytopenia and thrombosis (HITT or HIT type 2),
18. Suspected or known current alcohol or drug addiction,
19. History of active or previous autoimmune neurological disorders (e.g. multiple sclerosis, Guillain-Barre syndrome, transverse myelitis) (Lumbar palsy will not be an exclusion criterion),
20. Subjects with severe renal impairment or liver failure,
21. Acute respiratory disease (moderate or severe illness with or without fever). (Subjects may be screened again after acute condition has resolved).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy pregnant female subjects aged 18 - 45 years (including both groups)
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Incidence of adverse events throughout the entire study from first and second dose vaccinations.
  Incidence of obstetric, fetal, and neonatal adverse events of TURKOVAC vaccine.

SECONDARY OUTCOMES:
Neutralizing Antibodies and Pseudo-Neutralizing Antibodies | On days 0, 28±2 (for all subjects) 48±5, 84±5 ve 168±10 (for 50% of all subjects)
  The change in the amount of SARS-CoV 2 neutralizing antibodies and pseudo-neutralizing Antibodies in the 28th day compared to the baseline is 2 times and more.
SARS-CoV2 anti-spike protein immunoglobulin G | On days 0, 28±2 (for all subjects) 48±5, 84±5 ve 168±10 (for 50% of all subjects)
  The change in the amount of SARS-CoV2 anti-spike protein immunoglobulin G in the 28th day compared to the baseline is 2 times and more.
T-Cell | On the 28th day
  IL-2, TNF-alpha, and IFN-gamma levels in T cells changed by 2 times and more on day 28 compared to baseline.
Protection Rate of TURKOVAC | 24 hours (subjects with at least 1 symptom within 24 hours) and at least 14 days after the TURKOVAC vaccination dose.
  Protection rate of the TURKOVAC vaccine against COVID-19 in subjects with a positive real time-polymerase chain reaction (RT-PCR) test at least 14 days after the TURKOVAC vaccination and showing at least 1 symptom within 24 hours.
The antibody Level in the Cord Blood | Between Visit 0 (-1 or 0. day) Visit 4 (168 day ±10) (At the time of birth)
  The antibody level in the cord blood
Antibody Persistence | 6 months and 12 months after vaccination.
  Antibody persistence in mothers at 6 months and 12 months post-vaccination during pregnancy.
Incidence of Adverse Reactions | 7 to 14 days after vaccination.
  Incidence of adverse reactions in all subjects 7 to 14 days after vaccination.
Incidence of Serious Adverse Events (SAE) | Up to day 365 after vaccination.
  Incidence of Serious Adverse Events (SAE) in all subjects up to day 365 after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Moraloğlu Tekin, Prof., Principal Investigator — Faculty Member
Locations (1):
- T.R. Ministry of Health Ankara City Hospital, Gynecology and Obstetrics Hospital, Ankara, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar A, Singh R, Kaur J, Pandey S, Sharma V, Thakur L, Sati S, Mani S, Asthana S, Sharma TK, Chaudhuri S, Bhattacharyya S, Kumar N. Wuhan to World: The COVID-19 Pandemic. Front Cell Infect Microbiol. 2021 Mar 30;11:596201. doi: 10.3389/fcimb.2021.596201. eCollection 2021. PMID 33859951
- [Background] Pavel STI, Yetiskin H, Aydin G, Holyavkin C, Uygut MA, Dursun ZB, Celik I, Cevik C, Ozdarendeli A. Isolation and characterization of severe acute respiratory syndrome coronavirus 2 in Turkey. PLoS One. 2020 Sep 16;15(9):e0238614. doi: 10.1371/journal.pone.0238614. eCollection 2020. PMID 32936826
- [Background] Limaye MA, Roman AS, Trostle ME, Venkatesh P, Lantigua Martinez M, Brubaker SG, Chervenak J, Wei LS, Sahani P, Grossman TB, Meyer JA, Penfield CA. Predictors of severe and critical disease in pregnant women with SARS-CoV-2. J Matern Fetal Neonatal Med. 2022 Dec;35(25):7536-7540. doi: 10.1080/14767058.2021.1951216. Epub 2021 Sep 1. PMID 34470122
- [Background] Adhikari EH, Spong CY. COVID-19 Vaccination in Pregnant and Lactating Women. JAMA. 2021 Mar 16;325(11):1039-1040. doi: 10.1001/jama.2021.1658. No abstract available. PMID 33555297
- [Background] Goncu Ayhan S, Oluklu D, Atalay A, Menekse Beser D, Tanacan A, Moraloglu Tekin O, Sahin D. COVID-19 vaccine acceptance in pregnant women. Int J Gynaecol Obstet. 2021 Aug;154(2):291-296. doi: 10.1002/ijgo.13713. Epub 2021 May 1. PMID 33872386